CLINICAL TRIAL: NCT02234284
Title: Health Coaching to Reduce Disparities for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Aides in Respiration Health Coaching for COPD
Acronym: AIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PCORI AD-1306-03900
Record Dates: First submitted 2014-08-12; First posted 2014-09-09 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease; Health Coaching; Health Disparities; Self-management; Chronic Disease Model
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Coaching (Experimental): Patients randomized to the health coaching intervention would work with a trained health coach who would provide patient education self-management support, use action planning to help patient make changes to reach goals, as well as help coordinate patient care between the primary care provider and pulmonary specialist, identify gaps in care, and help patient access needed services
  Interventions: Behavioral: Health Coaching
- Usual care (No Intervention): Usual care was chosen as the comparison group to provide maximum generalizability of the study, as usual care is the practical alternative for the target population. Usual care includes patient education classes, smoking cessation classes, psychosocial medicine and nutritional counseling.

INTERVENTIONS:
Behavioral: Health Coaching — Patient COPD education; Correct use of inhalers and nebulizers; Red flags and when to seek medical care; Dyspnea management; Patient decision making and action plans around, exercise, smoking cessation; nutrition, exacerbations; Ensuring appropriate preventive services (pneumovax, flu); Depression screening; Reinforcing clinician education and use of treatment guidelines by primary care providers; Identifying gaps in care, areas where care not in line with care plan; Facilitating communication between patients, pulmonary specialists and primary care providers; Connecting with community resources; Access to psychosocial services; Working with pulmonary specialist to provide recommended exercise program; Working with patient family members and caregivers.
  Arms: Health Coaching

SUMMARY:
This study examined whether health coaches can improve the management of chronic obstructive pulmonary disease (COPD) in a population of vulnerable patients cared for in 'safety-net' clinics. The study is designed as a randomized controlled trial for patients with moderate to severe COPD. Patients were randomized into a health coaching group and a usual care group. Those in the health coaching group received 9 months of active health coaching. Outcome variables were measured at baseline and after 9 months

DETAILED DESCRIPTION:
Health coaching is a promising model for improving evidence-based care for patients with COPD which had not been evaluated at the time the current study began in 2014. Health coaching by health workers or peers trained as coaches, has emerged as an effective model to improve these management domains for children with asthma and adults with diabetes, and hypertension receiving care in urban safety-net clinics. The role of the health coach includes many of the activities also provided by patient navigators, patient educators, and community health workers. Health coaching is a patient-centered model that recognizes that that people living with chronic disease are the primary decision-makers in their care; it is a tailored approach that builds on the strengths and expertise of patients and helps to ensure that they have the knowledge and skills to be active participants within the medical encounter and to effectively manage their conditions. Incorporating health coaches into care delivery fits well with the of integrated care model recommended by the American Thoracic Society which is based on the Chronic Care Mode. Health coaching can work on several components of the Chronic Care Model as it applies to COPD to enhance the effectiveness of care delivery and promote patient goals. Health coaches provide decision support by helping execute customized care plans jointly developed by patients and providers. Coaches track care targets and conduct 'gap analysis' to identify areas which are sub-optimal. Coaches also help patients to get the support they need by facilitating access to community, clinic, and specialist support, improving communication between patients and providers, working with patients to set goals and develop action plans to reach those goals. The goal of our study was to evaluate the effectiveness of a health coach model for improving outcomes for low-income urban patients with COPD. We conducted a randomized trial comparing 9 months of health coaching plus usual care (health coached arm) to usual care (usual care arm) alone for patients with moderate to severe COPD cared for at 7 federally qualified health centers (FQHCs). The specific aims of the study were:

Specific Aim 1. To compare disease specific quality of life for patients randomized to receive 9 months of health coaching plus usual care to those randomized to usual care alone. Our hypothesis was that mean quality of life, assessed by the Chronic Respiratory Disease Questionnaire total score and dyspnea domain score at 9 months, would be greater in patients in the health-coached arm when tested against the null hypothesis of no difference between health-coached and usual care patients.

Specific Aim 2. To compare the number of exacerbations of COPD experienced by patients in the health coached arm to those in the usual care arm during the 9 month period starting at enrollment. COPD exacerbation was defined as an emergency department visit or hospitalization for COPD-related diagnosis or the outpatient prescription of oral steroids for COPD-related diagnosis. Our hypothesis was patients in the health-coached arm would experience fewer exacerbations when tested against the null hypothesis of no difference between health-coached and usual care patients.

Specific Aim 3. To compare exercise capacity at 9 months for patients in the health-coached arm to those in the usual care arm. Our hypothesis was that patients in the health-coached arm would have greater exercises capacity as measured by the 6-minute Walk Test when tested against the null hypothesis of no difference between health-coached and usual care patients.

Specific Aim 4. To compare self-efficacy for management of their COPD for health-coached versus usual care patients at 9 months. Our hypothesis was that mean self-efficacy, as measured by Stanford Chronic Disease Self-Efficacy Scale would be greater in patients in the health coached arm when tested against the null hypothesis of no difference in self-efficacy between health-coached and usual care patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient at one of the participating primary care clinics (at least 1 visit in past 12 months)
* Age 40 and older
* Speaking English or Spanish
* Plan to continue to be seen at current clinic and to not leave the area for >2 months anytime in the next 9 months or to be absent at 9 or 15 months
* COPD defined as ever having had a post-bronchodilator Forced Expiratory Volume in 1 second/Forced Vital Capacity (FEV1/FVC) <.70 of FEV1/FVC of .70 to .74 and diagnosis of COPD by the study pulmonologist
* Willingness to attempt spirometry
* At least moderate COPD, defined as at least one of the following:

  * Ever Forced Expiratory Volume in 1 second (FEV1) < 80% predicted
  * 1 or more emergency department (ED) visit for COPD exacerbation in past 12 months
  * 1 or more hospital stays for COPD exacerbation in past 12 months
  * 1 or more prescriptions for oral prednisone for a COPD exacerbation in past 12 months
  * Ever on home oxygen therapy
  * Ever outpatient percutaneous oxygen saturation of </=88%
  * Ever outpatient partial pressure of oxygen (ppO2) by arterial blood gas (ABG) of </=55mm Hg
  * At least 3 outpatient visits for COPD in past 12 months AND (a current COPD Assessment Test (CAT) score of >/=10 OR an modified Medical Research Council (mMRC) score of >/=2).
  * Currently using tiotropium inhaler or combination inhaled corticosteroid and long-acting beta agonist

Exclusion Criteria:

* Unable to participate in the study due to mental or physical impairment
* Severe or terminal illness that precludes focus on COPD
* No phone

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Thom, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Departmen of Public Health Community Clinics, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang B, Willard-Grace R, De Vore D, Wolf J, Chirinos C, Tsao S, Hessler D, Su G, Thom DH. Health coaching to improve self-management and quality of life for low income patients with chronic obstructive pulmonary disease (COPD): protocol for a randomized controlled trial. BMC Pulm Med. 2017 Jun 9;17(1):90. doi: 10.1186/s12890-017-0433-3. PMID 28599636
- [Background] Huang B, De Vore D, Chirinos C, Wolf J, Low D, Willard-Grace R, Tsao S, Garvey C, Donesky D, Su G, Thom DH. Strategies for recruitment and retention of underrepresented populations with chronic obstructive pulmonary disease for a clinical trial. BMC Med Res Methodol. 2019 Feb 21;19(1):39. doi: 10.1186/s12874-019-0679-y. PMID 30791871
- [Result] Thom DH, Willard-Grace R, Tsao S, Hessler D, Huang B, DeVore D, Chirinos C, Wolf J, Donesky D, Garvey C, Su G. Randomized Controlled Trial of Health Coaching for Vulnerable Patients with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2018 Oct;15(10):1159-1168. doi: 10.1513/AnnalsATS.201806-365OC. PMID 30130430
- [Derived] Willard-Grace R, Chirinos C, Wolf J, DeVore D, Huang B, Hessler D, Tsao S, Su G, Thom DH. Lay Health Coaching to Increase Appropriate Inhaler Use in COPD: A Randomized Controlled Trial. Ann Fam Med. 2020 Jan;18(1):5-14. doi: 10.1370/afm.2461. PMID 31937527

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Coaching: Major health coach activities:
  Patient COPD education; Correct use of inhalers and nebulizers; Identifying red flags and when to seek medical care; Dyspnea management; Patient decision making and action plans around, exercise, smoking cessation, nutrition, exacerbations; Ensuring appropriate preventive services (pneumovax, flu); Depression screening; Reinforcing clinician education and use of treatment guidelines by primary care providers; Helping patient obtain prescriptions; Identifying gaps in care, areas where care not in line with care plan; Helping patients to make and keep appointments and obtain needed testing; Facilitating communication between patients, pulmonary specialists and primary care providers; Connecting with community resources; Helping to access to psychosocial services as needed; Conducting exercise capacity assessment and working with pulmonary specialist to provide recommended exercise program; Working with patient family members a
- Usual Care: Usual care includes access to specialist consultation via referral by the primary care clinician, access to patient education classes, smoking cessation classes, psychosocial medicine and nutritional counseling.
Period: Overall Study
Arm/Group | Health Coaching | Usual Care
Started | 100 | 92
Completed | 75 | 83
Not Completed | 25 | 9
Not completed — Death | 4 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 20 | 7

BASELINE CHARACTERISTICS:
Groups:
- Health Coaching: Coaching activities: Patient COPD education Correct use of inhalers and nebulizers Red flags and when to seek medical care Dyspnea management Use of oxygen Patient decision making and action plans around, exercise, smoking cessation, nutrition, exacerbations Ensuring appropriate preventive services (pneumovax, flu) Depression screening Reinforcing clinician education and use of treatment guidelines by primary care providers Helping patient obtain prescriptions Identifying gaps in care, areas where care not in line with care plan Helping patients to make and keep appointments and obtain needed testing Facilitating communication between patients, pulmonary specialists and primary care providers Connecting with community resources Access to psychosocial services Conducting exercise capacity assessment and working with pulmonary specialist to provide recommended exercise program Working with patient family members and caregivers
- Total: Total of all reporting groups
Arm/Group | Health Coaching | Usual Care | Total
Number analyzed (Participants) | 100 | 92 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 54 | 121
  >=65 years | 33 | 38 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.0) | 61.9 (7.1) | 61.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 67 | 59 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 19 | 32
  Not Hispanic or Latino | 87 | 73 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 53 | 56 | 109
  White | 29 | 12 | 41
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 12 | 13 | 25
Short Form Chronic Respiratory Disease Questionnaire (CRQ-SF) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Chronic Respiratory Disease Questionnaire assesses disease-related quality of in 4 domains (dyspnea, fatigue, physical function and mastery). The 8-item Short Form version has been validated against the original full version. Each item is answered on a 7-point response scale where a higher score indicates a higher quality of life. The measure is scored as the mean response score (range 1 to 7) for each domain and for the total score, with the higher score indicating higher quality of life.
  units on a scale | 4.24 (1.22) | 4.28 (1.23) | 4.26 (1.22)
Dyspnea Domain Score of the Short Form of the Chronic Respiratory Disease Questionnaire (CRQ-SF) [Mean (Standard Deviation); unit: units on a scale] — The CRQ-SF is the short-form version of the original Chronic Respiratory Disease Questionnaire. The CRQ-SF has a total of 8 items asking about the frequency of COPD-related symptoms in 4 domains (2 questions per domain): Dyspnea, Fatigue, Emotional Function and Mastery. Each item is answered on a 7-point Likert-type scale with 1=none of the time and 7=all of the time. The dyspnea score is reported as the mean of the two items asking about shortness of breath. Mean scores range for 1 to 7, with a higher score indicating a worse quality of life related to dyspnea. Population: missing data
  units on a scale
    number analyzed (Participants) | 99 | 91 | 190
    (all) | 4.39 (1.46) | 4.63 (1.45) | 4.51 (1.46)
Rate of COPD exacerbations [Mean (Standard Deviation); unit: events per person year] — A COPD exacerbation was defined as a COPD-related emergency department visit or hospitalization, or the outpatient prescription of oral steroids and/or antibiotic for COPD-related diagnosis, as documented in the medical record. The rate of COPD exacerbation was calculated as the mean number of exacerbations per participant per year.
  events per person year | 0.95 (1.57) | 0.92 (1.34) | 0.94 (1.46)
Exercise capacity (6-Minute Walk Test) [Mean (Standard Deviation); unit: meters] — Distance walked, in meters, over 6 minutes. Higher number indicates greater exercise capacity. Population: Some participants were unable to do this test
  meters
    number analyzed (Participants) | 71 | 65 | 136
    (all) | 305 (83.1) | 292 (77.5) | 299 (80.4)
Self-efficacy to Manage Chronic Disease Scale [Mean (Standard Deviation); unit: units on a scale] — The Self-efficacy to Manage Chronic Disease Scale is a validated measure of of patient self-efficacy for managing a specific chronic disease (in this case, COPD). The Self-efficacy to Manage Chronic Disease Scale has 6 items asking about patients' self-confidence dealing with 6 aspects off self-management. Each item is answered on a scale of 1 to 10 with 1="not at all confident" and 10='totally confident". The score is the mean of all 10-items. Mean scores range for 1 to 10, with a higher score indicating greater self-efficacy for managing COPD.
  units on a scale | 6.36 (2.23) | 6.45 (2.11) | 6.40 (2.17)
Short version of the Patient Assessment of Quality of Care (PACIC) [Mean (Standard Deviation); unit: units on a scale] — Patient Assessment of Chronic Illness Care (PACIC) is a patient reported measure of having received services recommended by Chronic Care Model. The short version of the PACIC has 11 items asking the patient the proportion of time he or she received a specific service. Each item is answered on a 5-point Likert-type scale with 1=None of the time and 5=Always. The total score is the mean of all 11-items. Mean scores range for 1 to 5, with a higher score indicating higher quality of care. Population: missing data
  units on a scale
    number analyzed (Participants) | 93 | 85 | 178
    (all) | 3.58 (.98) | 3.29 (1.20) | 3.45 (1.10)
COPD Symptoms (COPD Assessment Test) [Mean (Standard Deviation); unit: units on a scale] — The COPD Assessment Test (CAT) is an 8-item measure of severity of COPD symptoms, with responses from 1 to 5 . It is scored as the sum of item scores, with a range from 8 to 40, with a higher score indicating greater level of symptoms.
  units on a scale | 20.6 (8.34) | 20.9 (7.41) | 20.7 (7.89)
Lung Function (FEV1 % predicted) [Mean (Standard Deviation); unit: percent of predicted] — Volume of air exhaled, using maximal force, over 1 second, divided by the volume expected for health person of same age and gender. Larger volume indicates better lung function. Population: We were not able to obtain spirometry on all patients due to contraindications or technical limitations
  percent of predicted
    number analyzed (Participants) | 79 | 73 | 152
    (all) | 0.55 (0.19) | 0.60 (0.20) | 0.58 (0.20)
Proportion (%) of Participants reporting Current Cigarette Use [Count of Participants; unit: Participants] — Current cigarette use is defined as any use in the past 30 days. Population: missing data
  Participants
    number analyzed (Participants) | 99 | 85 | 184
    (all) | 54 | 45 | 99
Proportion (%) of Participants Demonstrating Adequate Inhaler Use [Count of Participants; unit: Participants] — Observational measure using a check list to document mistakes in using inhalers. Adequate use defined as correctly performing all necessary steps for every inhaler used. Definition of necessary steps varies by type of inhaler. Population: Some participants did not have inhalers prescribed at baseline
  Participants
    number analyzed (Participants) | 95 | 83 | 178
    (all) | 12 | 5 | 17
COPD-related function (Bed days in past 4 weeks due to respiratory problems) [Mean (Standard Deviation); unit: days] — Number of days in past 4 weeks where COPD keep participant in bed all or most of the day. Population: missing data
  days
    number analyzed (Participants) | 99 | 90 | 189
    (all) | 2.75 (6.44) | 3.86 (6.86) | 3.28 (6.65)
Proportion (%) of Participants With Correct Answer to Knowledge Question 1 [Count of Participants; unit: Participants] — Okay to get short of breath while exercising (correct answer is yes) Population: question not answered by 2 participants
  Participants
    number analyzed (Participants) | 100 | 90 | 190
    (all) | 75 | 64 | 139
Proportion (%) of Participants With Correct Answer to Knowledge Question 2 [Count of Participants; unit: Participants] — Beneficial to stop smoking (correct answer is yes) Population: question not answered by 2 participants
  Participants
    number analyzed (Participants) | 100 | 90 | 190
    (all) | 83 | 75 | 158
Proportion (%) of Participants With Correct Answer to Knowledge Question 3 [Count of Participants; unit: Participants] — Okay to be on oxygen long term (correct answer) Population: not answered by 3 participants
  Participants
    number analyzed (Participants) | 99 | 89 | 188
    (all) | 67 | 50 | 117
Proportion (%) of Participants With Correct Answer to Knowledge Question 4 [Count of Participants; unit: Participants] — Smoking does not help breathing (correct answer) Population: Question not answered by 3 participants
  Participants
    number analyzed (Participants) | 99 | 90 | 189
    (all) | 96 | 85 | 181
Rate of all outpatient visits [Mean (Standard Deviation); unit: visits per patient per year] — Number of visits to primary care provider, pulmonary specialist or urgent care, per patient per year, over 12 months prior to enrollment
  visits per patient per year | 6.62 (5.43) | 6.53 (4.08) | 6.58 (4.82)
Rate of emergency department (ED) visits for COPD [Mean (Standard Deviation); unit: visits per patient per year] — Number of visits to emergency department for COPD exacerbation, per patient per year, over 12 months prior to enrollment
  visits per patient per year | 0.54 (1.26) | 0.62 (1.19) | 0.58 (1.23)
Rate of all ED visits not for COPD [Mean (Standard Deviation); unit: visits per patient per year] — Number of visits to emergency department not for a COPD exacerbation, per patient per year, over 12 months prior to enrollment
  visits per patient per year | 1.12 (2.52) | 0.62 (1.29) | 0.88 (2.03)
Rate of hospitalizations for COPD [Mean (Standard Deviation); unit: hospitalizations per patient per year] — Number of hospital admissions for COPD exacerbation, per patient per year, over 12 months prior to enrollment
  hospitalizations per patient per year | 0.13 (0.39) | 0.34 (0.77) | 0.23 (0.61)
Rate of hospitalizations not for COPD [Mean (Standard Deviation); unit: hospitalizations per patient per year] — Number of hospital admissions not for a COPD exacerbation, per patient per year, over 12 months prior to enrollment
  hospitalizations per patient per year | 0.21 (0.57) | 0.18 (0.44) | 0.20 (0.51)
Proportion (%) of participants receiving guideline-concordant medications for COPD [Count of Participants; unit: Participants] — Prescription of medications for COPD in concordance with the recommendations from the Global Initiative for Obstructive Lung Disease (GOLD) Guideline, based on classification categories of A, B C or D. Population: unable to determine GOLD classification for 2 patients (1 in each study arm)
  Participants
    number analyzed (Participants) | 99 | 91 | 190
    (all) | 72 | 63 | 135
Proportion (%) of Patients with a score of >/= 15 on the Patient Health Questionnaire 8 item version [Count of Participants; unit: Participants] — Patient Health Questionnaire (PHQ) 8 item version (without suicidality item) of the PHQ-9. The 8 items, which ask about the frequency of symptoms of depression, are answered on a likert-type scale from 0 to 3, with 0= 'not at all' and 3='nearly every day'. The total score ranges from 0 to 24, with a higher score indication more more severe depression symptoms. A score of >/= 15 indicates symptoms of at least moderate depression. Population: missing data on 1 participant
  Participants
    number analyzed (Participants) | 100 | 91 | 191
    (all) | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Short Form Chronic Respiratory Disease Questionnaire (CRQ-SF) Total Score
Description: The Chronic Respiratory Disease Questionnaire assesses disease-related quality of in 4 domains (dyspnea, fatigue, physical function and mastery). The 8-item Short Form version has been validated against the original full version. Each item is answered on a 7-point response scale where a higher score indicates a higher quality of life. The measure is scored as the mean response score (range 1 to 7) for each domain and for the total score, with the higher score indicating higher quality of life.
Time Frame: 9 months
Population: All participants who completed the CRQ-SF at 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Health Coaching: Health coaching included the following activities Patient COPD education; Correct use of inhalers and nebulizers; Red flags and when to seek medical care; Dyspnea management; Patient decision making and action plans around, exercise, smoking cessation, nutrition, exacerbations; Ensuring appropriate preventive services (pneumovax, flu); Depression screening; Reinforcing clinician education and use of treatment guidelines by primary care providers; Helping patient obtain prescriptions Identifying gaps in care, areas where care not in line with care plan;Helping patients to make and keep appointments and obtain needed testing; Facilitating communication between patients, pulmonary specialists and primary care providers; Connecting with community resources; Helping to access to psychosocial services ; Conducting exercise capacity assessment and working with pulmonary specialist to provide recommended exercise program ; Working with patient family members and caregivers
- Usual Care: Patients the usual care arm could be referred to a specialist by their primary care clinician and had access to education classes, smoking cessation classes, psychosocial medicine and nutritional counseling.
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 75 | 83
units on a scale | 4.58 (1.25) | 4.43 (1.28)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; Outcomes were compared by group assignment using generalized linear models (GLMs) with a normal distribution for continuous outcomes), Poisson distribution for count outcomes (e.g. exacerbations and hospitalizations), and binomial distribution for binary outcomes. In all models, baseline levels of the outcome were entered as a predictor and follow-up levels as the dependent variable, with use of a robust standard error to account for clustering; Test type: Superiority; p = .35, Mixed Models Analysis; Outcomes were by group assignment (intention to treat) using generalized linear models adjusted for baseline levels of variable and clustering; Mean Difference (Final Values) = .14, 95% CI 2-sided [-.15 to .43] — Value is for mean score of participants in Health Coached arm minus mean score in Usual Care, adjusted for baseline values and for clustering

2. Primary Outcome: Dyspnea Domain Score of the Short Form of the Chronic Respiratory Disease Questionnaire (CRQ-SF)
Description: The CRQ-SF is the short-form version of the original Chronic Respiratory Disease Questionnaire. The CRQ-SF has a total of 8 items asking about the frequency of COPD-related symptoms in 4 domains (2 questions per domain): Dyspnea, Fatigue, Emotional Function and Mastery. Each item is answered on a 7-point Likert-type scale with 1=none of the time and 7=all of the time. The dyspnea score is reported as the mean of the two items asking about shortness of breath. Mean scores range for 1 to 7, with a higher score indicating a worse quality of life related to dyspnea.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 75 | 83
units on a scale | 4.98 (1.39) | 4.78 (1.49)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .20, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = .26, 95% CI 2-sided [-.13 to .65] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Rate of COPD Exacerbations Per Year
Description: A COPD exacerbation was defined as a COPD-related emergency department visit or hospitalization, or the outpatient prescription of oral steroids and/or antibiotic for COPD-related diagnosis, as documented in the medical record over the 9 month trial period. The rate of COPD exacerbation was calculated as the mean number of exacerbations per participant per year.
Time Frame: Over 9 month study period
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 100 | 92
events | 1.17 (1.87) | 1.44 (2.16)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .13, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.21, 95% CI 2-sided [-0.49 to 0.07] — Value is for rate of exacerbations for participants in Health Coached arm minus rate for Usual Care, adjusted for baseline values and for clustering

4. Secondary Outcome: Exercise Capacity (6-minute Walk Test)
Description: Distance walked, in meters, over 6 minutes. Higher number indicates greater exercise capacity.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 37 | 42
Meters | 326 (68.3) | 311 (73.8)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .32, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.53, 95% CI 2-sided [-8.18 to 25.26]; Value is for mean distance (in meters) of participants in Health Coached arm minus mean distance in Usual Care, adjusted for baseline values and for clustering

5. Secondary Outcome: Self-efficacy to Manage Chronic Disease Scale
Description: The Self-efficacy to Manage Chronic Disease Scale is a validated measure of of patient self-efficacy for managing a specific chronic disease (in this case, COPD). The Self-efficacy to Manage Chronic Disease Scale has 6 items asking about patients' self-confidence dealing with 6 aspects off self-management. Each item is answered on a scale of 1 to 10 with 1="not at all confident" and 10='totally confident". The score is the mean of all 10-items. Mean scores range for 1 to 10, with a higher score indicating greater self-efficacy for managing COPD.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 73 | 83
units on a scale | 6.84 (2.01) | 6.50 (2.00)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .27, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .30, 95% CI 2-sided [-.23 to .83] — [estimate comment as in outcome 1, analysis 1]

6. Other Pre Specified Outcome: Short Version of the Patient Assessment of Quality of Care (PACIC)
Description: Patient Assessment of Chronic Illness Care (PACIC) is a patient reported measure of having received services recommended by Chronic Care Model. The short version of the PACIC has 11 items asking the patient the proportion of time he or she received a specific service. Each item is answered on a 5-point Likert-type scale with 1=None of the time and 5=Always. The total score is the mean of all 11-items. Mean scores range for 1 to 5, with a higher score indicating higher quality of care.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 72 | 72
units on a scale | 3.91 (0.95) | 3.44 (1.17)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .02, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = .38, 95% CI 2-sided [.07 to .68] — [estimate comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: COPD Assessment Test
Description: The COPD Assessment Test (CAT) is an 8-item measure of severity of COPD symptoms, with responses from 1 to 5 . It is scored as the sum of item scores, with a range from 8 to 40, with a higher score indicating greater level of symptoms.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Health Coaching: Health coaching included the following activities Patient COPD education; Correct use of inhalers and nebulizers; Red flags and when to seek medic al care; Dyspnea management; Patient decision making and action plans around, exercise, smoking cessation, nutrition, exacerbations; Ensuring appropriate preventive services (pneumovax, flu); Depression screening; Reinforcing clinician education and use of treatment guidelines by primary care providers; Helping patient obtain prescriptions Identifying gaps in care, areas where care not in line with care plan;Helping patients to make and keep appointments and obtain needed testing; Facilitating communication between patients, pulmonary specialists and primary care providers; Connecting with community resources; Helping to access to psychosocial services ; Conducting exercise capacity assessment and working with pulmonary specialist to provide recommended exercise program ; Working with patient family members and caregivers
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 74 | 83
units on a scale | 19.1 (8.80) | 20.2 (9.25)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .40, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-2.78 to 1.12] — [estimate comment as in outcome 1, analysis 1]

8. Other Pre Specified Outcome: Percent of Predicted Force Expiratory Volume at 1 Second (FEV1)
Description: Volume of air exhaled, using maximal force, over 1 second, divided by the volume expected for health person of same age and gender. Larger volume indicates better lung function.
Time Frame: 9 months
Population: Participants completing measurement of FEV1 % Predicted at 9 months
Measure: Mean (Standard Error); unit: Percent of predicted value
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 55 | 54
Percent of predicted value | 0.55 (0.20) | .59 (.21)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .98, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0, 95% CI 2-sided [-3 to 3] — Value is for mean percent predicted of participants in Health Coached arm minus mean percent predicted in Usual Care, adjusted for baseline values and for clustering

9. Other Pre Specified Outcome: Proportion (%) of Participants Reporting Current Cigarette Use
Description: Current cigarette use is defined as any use in the past 30 days.
Time Frame: 9 months
Population: Participants reporting smoking status at 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 77 | 81
Participants | 29 | 34
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .30, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.5, 95% CI 2-sided [-33.3 to 10.2] — Value is for proportion (%) of participants in Health Coached arm minus proportion in Usual Care, adjusted for baseline values and for clustering

10. Other Pre Specified Outcome: COPD-related Function (Bed Days Due to Respiratory Problems)
Description: Number of days in past 4 weeks where COPD keep participant in bed all or most of the day.
Time Frame: 9 months
Population: Participants reporting bed days at 9 monhts
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 74 | 83
Days | 2.15 (5.76) | 3.64 (6.81)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; Test type: Superiority; p = .29, Mixed Models Analysis; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-2.07 to 0.62] — Value is for mean number of days for participants in Health Coached arm minus mean score in Usual Care, adjusted for baseline values and for clustering

11. Other Pre Specified Outcome: Proportion (%) of Participants Demonstrating Adequate Inhaler Use
Description: Observational measure using a check list to document mistakes in using inhalers. Adequate use defined as correctly performing all necessary steps for every inhaler used. Definition of necessary steps varies by type of inhaler.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 70 | 77
Participants | 27 | 9
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 39.7, 95% CI 2-sided [19.6 to 59.8] — [estimate comment as in outcome 9, analysis 1]

12. Other Pre Specified Outcome: Proportion (%) of Participants With Correct Answer to Knowledge Question 1
Description: Okay to get short of breath while exercising
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 74 | 82
Participants | 54 | 56
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .38, Mixed Models Analysis; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-9.5 to 25.2] — Value is for proportion of participants in Health Coached arm minus proportion in Usual Care, adjusted for baseline values and for clustering

13. Other Pre Specified Outcome: Proportion (%) of Participants With Correct Answer to Knowledge Question 2
Description: beneficial to stop smoking
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 74 | 82
Participants | 67 | 73
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .73, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 2.0, 95% CI 2-sided [-9.4 to 13.4]

14. Other Pre Specified Outcome: Proportion (%) of Participants With Correct Answer to Knowledge Question 3
Description: Okay to be on oxygen for long period
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 74 | 82
Participants | 51 | 52
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .70, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-14.0 to 20.8] — [estimate comment as in outcome 9, analysis 1]

15. Other Pre Specified Outcome: Proportion (%) of Participants With Correct Answer to Knowledge Question 4
Description: Smoking does not help breathing
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 74 | 82
Participants | 72 | 80
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .97, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-5.5 to 5.3] — [estimate comment as in outcome 9, analysis 1]

16. Other Pre Specified Outcome: Rate of Outpatient Visits
Description: Number of outpatient visits per patient per year
Time Frame: Over 9 month study period
Measure: Mean (Standard Deviation); unit: visits per patient per year
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 100 | 92
visits per patient per year | 7.51 (5.64) | 6.83 (4.73)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .52, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-0.32 to 1.28] — Value is for rate of outpatient visits for participants in Health Coached arm minus rate for Usual Care, adjusted for baseline values and for clustering

17. Other Pre Specified Outcome: Rate of ED Visits for COPD
Description: Number of ED visits for COPD per patient per year over 9 month study period
Time Frame: Over 9 month study period
Measure: Mean (Standard Deviation); unit: Visits per patient per year
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 100 | 92
Visits per patient per year | 0.80 (1.63) | 0.89 (1.99)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .78, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.32 to 0.22] — Value is for rate of COPD-related ED visits for participants in Health Coached arm minus rate for Usual Care, adjusted for baseline values and for clustering

18. Other Pre Specified Outcome: Rate of ED Visits Not for COPD
Description: Number of visits to emergency department other than for COPD related reason per patient per year during 9 month study period
Time Frame: Over 9 month study period
Measure: Mean (Standard Deviation); unit: Visits per patient per year
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 100 | 92
Visits per patient per year | 0.98 (1.89) | 0.83 (2.33)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .80, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.56 to 0.40] — Value is for rate of non-COPD-related ED visits for participants in Health Coached arm minus rate for Usual Care, adjusted for baseline values and for clustering

19. Other Pre Specified Outcome: Rate of Hospitalization for COPD
Description: Number of hospitalizations for COPD per patient per year over 9 month study period
Time Frame: Over 9 month study period
Measure: Mean (Standard Deviation); unit: Hospitalizations per patient per year
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 100 | 92
Hospitalizations per patient per year | 0.27 (0.77) | 0.52 (1.25)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .35, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.32 to 0.06] — Value is for rate of COPD-related hospital visits for participants in Health Coached arm minus rate for Usual Care, adjusted for baseline values and for clustering

20. Other Pre Specified Outcome: Rate of Hospitalizations Not for COPD
Description: Number of hospitalizations other than for COPD per patient per year during 9 month study period
Time Frame: Over 9 month study period
Measure: Mean (Standard Deviation); unit: Hospitalizations per patient per year
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 100 | 92
Hospitalizations per patient per year | 0.16 (0.58) | 0.21 (0.81)
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .37, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.20 to 0.04] — Value is for rate of non-COPD-related hospitalizations for participants in Health Coached arm minus rate for Usual Care, adjusted for baseline values and for clustering

21. Post Hoc Outcome: Proportion (%) of Patients With a Score of >/= 15 on the Patient Health Questionnaire 8 Item Version
Description: Patient Health Questionnaire (PHQ) 8 item version (without suicidality item) of the PHQ-9. The 8 items, which ask about the frequency of symptoms of depression, are answered on a likert-type scale from 0 to 3, with 0= 'not at all' and 3='nearly every day'. The total score ranges from 0 to 24, with a higher score indication more more severe depression symptoms. A score of >/= 15 indicates symptoms of at least moderate depression.
Time Frame: 9 month study period
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 72 | 82
Participants | 4 | 16
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .01, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; difference in proportion = -18.9, 95% CI 2-sided [-33.1 to -4.8] — [estimate comment as in outcome 9, analysis 1]

22. Post Hoc Outcome: Proportion (%) of Participants Receiving Guideline-concordant Medications for COPD.
Description: Prescription of medications for COPD in concordance with the recommendations from the Global Initiative for Obstructive Lung Disease (GOLD) Guideline, based on classification categories of A, B C or D.
Time Frame: 9 month study period
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Usual Care
Number analyzed (Participants) | 99 | 91
Participants | 91 | 72
Statistical Analysis 1: Comparison: Health Coaching vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .01, Mixed Models Analysis; Mean Difference (Final Values) = 14.6, 95% CI 2-sided [3.3 to 25.9] — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Health Coaching: Health coaching included the following activities Patient COPD education; Correct use of inhalers and nebulizers; Red flags and when to seek medical care; Dyspnea management; Patient decision making and action plans around, exercise, smoking cessation, nutrition, exacerbations; Ensuring appropriate preventive services (pneumovax, flu); Depression screening; Reinforcing clinician education and use of treatment guidelines by primary care providers; Helping patient obtain prescriptions Identifying gaps in care, areas where care not in line with care plan;Helping patients to make and keep appointments and obtain needed testing; Facilitating communication between patients, pulmonary specialists and primary care providers; Connecting with community resources; Helping to access to psychosocial services; Conducting exercise capacity assessment and working with pulmonary specialist to provide recommended exercise program; Working with patient family members and caregivers
Arm/Group | Health Coaching | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/100 | 2/92
Serious Adverse Events (participants affected / at risk) | 23/100 | 25/92
Other Adverse Events (participants affected / at risk) | 48/100 | 43/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Coaching (N=100) | Usual Care (N=92)
Hospitalization for COPD related diagnosis (Respiratory, thoracic and mediastinal disorders) | 14 (20) | 20 (35)
Hospitalization for other than COPD related diagnosis (General disorders) | 9 (12) | 8 (14)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Coaching (N=100) | Usual Care (N=92)
ED visit for COPD related diagnosis (Respiratory, thoracic and mediastinal disorders) | 29 (59) | 28 (57)
ED visit for non-COPD related diagnosis (General disorders) | 33 (73) | 25 (57)

LIMITATIONS AND CAVEATS:
Target sample size was reduced from 250 to 190 due difficulties with recruitment.

The outcome of medication adherence, measured by the Morisky Medication Adherence Scale, was deleted because we did not realized it required a license.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-09-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02234284/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02234284/SAP_001.pdf